CLINICAL TRIAL: NCT04972799
Title: AUTOGRAFI : Evaluation of the Efficacy and Safety of Autologous Fat Injection Into the Intersphincter Space in Fecal Incontinence: a Randomized, Placebo-controlled, Cross-over, Double-blind Trial
Brief Title: Evaluation of the Efficacy and Safety of Autologous Fat Injection Into the Intersphincter Space in Fecal Incontinence: a Randomized, Placebo-controlled, Cross-over, Double-blind Trial
Acronym: AUTOGRAFI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 35RC19_9798_AUTOGRAFI; 2020-A01890-39 (Other: N° IDRCB)
Record Dates: First submitted 2021-07-12; First posted 2021-07-22 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Fecal Incontinence
Keywords: Autograft
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment/Placebo (Experimental): treatment sequence at day 0 and placebo sequence at 6 months
  Interventions: Other: injection of autologous fat at Day 0 and injection of saline at 6 months
- Placebo/Treatment (Experimental): placebo sequence at day 0 and treatment sequence at 6 months
  Interventions: Other: injection of saline at Day 0 and injection of autologous fat at 6 months

INTERVENTIONS:
Other: injection of autologous fat at Day 0 and injection of saline at 6 months — injection into the intersphincter space
  Arms: Treatment/Placebo
Other: injection of saline at Day 0 and injection of autologous fat at 6 months — injection into the intersphincter space
  Arms: Placebo/Treatment

SUMMARY:
Fecal incontinence is frequent and has a significant impact on the quality of life of individuals. Its therapeutic management is based primarily on transit regulation and rehabilitation and secondarily on neuromodulation of the sacral roots. However, this strategy is insufficient in more than one patient out of three. The patient and the clinician are often at a loss and the therapeutic possibilities are limited to the use of evacuating enemas and/or a colostomy.

The practice of autologous fat injections was initially developed in plastic surgery. The studies that have evaluated the efficacy of autologous fat injections in fecal incontinence in men are preliminary and old isolated observations. However, they have shown an improvement in episodes of fecal incontinence and in sphincter parameters. In the field of proctology and autologous fat injections, 2 recent small open studies have evaluated the efficacy and morbidity of this therapy in the treatment of anal fistulas related to Crohn's disease.

The primary hypothesis of the work is that autografting adipose tissue into the intersphincteric space can decrease episodes of fecal incontinence in patients with severe fecal incontinence due to sphincter failure. The secondary hypotheses are that autograft of adipose tissue in the intersphincter space improves resting anal pressures, is a well-tolerated technique for patients, and may improve their quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. severe fecal incontinence characterized by at least one episode of weekly fecal incontinence
3. failed rehabilitation and dietary management strategies
4. who have failed/contraindicated/refused sacral root neuromodulation (in the indication of fecal incontinence)
5. having, for women of childbearing age, effective contraception throughout the study
6. having given free, informed and written consent

Exclusion Criteria:

1. unable or unwilling to undergo follow-up or symptomatic evaluation
2. contraindication to general anesthesia
3. contraindication to metronidazole (hypersensitivity and wheat allergy)
4. significant pelvic static disorder
5. active anal suppuration
6. anal stenosis
7. externalized rectal prolapse
8. chronic inflammatory bowel disease (Crohn's disease, ulcerative colitis)
9. on anticoagulants or antiaggregants
10. history of anal or rectal neoplasia
11. coagulation anomaly, curative anticoagulation
12. history of rectal surgery
13. history of pelvic radiotherapy
14. previous treatment with inert materials (hyaluronic acid, biosilicones, coaptitis) in the 5 years preceding inclusion
15. allergy to lidocaine or contraindication to adrenaline
16. protected person (adult subject to legal protection (safeguard of justice, curatorship, guardianship), person deprived of liberty, pregnant or breast-feeding woman, minor)
17. participating in another interventional trial concurrently
18. not covered by a social security system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-10-19 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Number of fecal incontinence events | 3 months
  Change from baseline in number of fecal incontinence events at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Brochard Charlène, Principal Investigator — CHU Rennes
Locations (3):
- France (3):
  - CHU Angers, Angers
  - CHU Nantes, Nantes
  - CHU Rennes, Rennes

IPD SHARING:
Plan to Share IPD: No